CLINICAL TRIAL: NCT03592693
Title: A Randomized, Double Blind, Placebo-Controlled Trial to Investigate the Effect of Vitamin C, Hydrocortisone and Thiamine on the Outcome of Patients with Septic Shock
Brief Title: Vitamin C, Hydrocortisone and Thiamine for Septic Shock
Acronym: CORVICTES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low rate of enrollment; publication of relevant results by other groups
Sponsor: University of Athens (Other)
Collaborators: General Hospital of Nikaia "Saint Panteleimon" (Other); Naval Hospital, Athens (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Associate Professor of Intensive Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 236-16-10-2017
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Shock, Septic
Keywords: Shock, Septic; Vitamin C; Hydrocortisone
MeSH Terms: conditions — Shock, Septic | interventions — PACEBO protocol

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, parallel group, placebo-controlled [Vitamin c plus hydrocortisone or placebo plus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators performing the follow-up, and care providers will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin-Steroid (Experimental): "Combined Vitamin C and Stress-Dose Hydrocortisone": Patients with septic shock treated with 1500 mg Vitamin C every 6 hours for 4 days after randomization, and stress-dose hydrocortisone for 4 days (250 mg on day 1; and 200 mg on days 2, 3, and 4) after randomization.
  Interventions: Drug: Combined Vitamin C and Stress-Dose Hydrocortisone
- Control (Placebo Comparator): "Placebo plus placebo:" Patients with septic shock treated with placebo (corresponding to Vitamin C) and placebo (corresponding to hydrocortisone) for 4 days after randomization.
  Interventions: Drug: Placebo plus placebo

INTERVENTIONS:
Drug: Combined Vitamin C and Stress-Dose Hydrocortisone — Treatment of septic shock with vitamin C and stress-dose hydrocortisone aimed at the attenuation of the systemic inflammatory response and the improvement of vasopressor responsiveness.
  Other Names: Vitamin-Steroid
  Arms: Vitamin-Steroid
Drug: Placebo plus placebo — Treatment of septic shock with placebo (corresponding to Vitamin C) and placebo (corresponding to hydrocortisone).
  Other Names: Pacebo
  Arms: Control

SUMMARY:
Prior data has shown that both corticosteroids and vitamin C reduce the activation of nuclear factor ƘB (NFƘB), thereby ultimately attenuating the systemic inflammatory response to sepsis/septic shock and augmenting the responsiveness to vasopressors. Therefore, the current investigators hypothesized that the combined use of vitamin C and stress-dose hydrocortisone may improve the outcomes of patients with septic shock. The investigators intend to perform a randomized, multicenter, parallel group, double-blind, placebo-controlled trial of vitamin C plus stress-dose hydrocortisone or placebo plus placebo for a total of four days after randomization of patients fulfilling the current consensus criteria for septic shock. The primary outcome will be hospital mortality, whereas the scondary outcomes will include 60-day, 28-day mortality, time to vasopressor cessation, procalcitonin clearance and change in the Sequential Organ Failure Assessment score over the first 4 days after randomization, neurologic failure-free days, and length of stay in the intensive care unit (ICU) and the hospital. Target enrollment will be 400 patients.

DETAILED DESCRIPTION:
Background and Significance:

The global burden of sepsis is substantial with an estimated 15 to 19 million cases per year; the vast majority of these cases occur in low income countries. With more timely diagnosis and improvement in supportive care the 28-day mortality from sepsis in high income countries has declined to about 25%, however, the mortality from septic shock remains as high as 45%. Moreover, the mortality from sepsis and septic shock in low income countries is reported to be as high as 60%. Over the last 3 decades over 100 phase II and phase III clinical trials have been performed testing various novel pharmacologic agents and therapeutic interventions in an attempt to improve the outcome of patients with sepsis and septic shock; all of these studies have failed to show an improvement in patient outcomes. A large body of experimental data has demonstrated that both corticosteroids and intravenous vitamin C reduce activation of nuclear factor ƘB (NFƘB) and attenuatethe release of pro-inflammatory mediators, reduce the endothelial injury characteristic of sepsis (thereby reducing endothelial permeability and improving macrocirculatory flow), augment the release of endogenous catecholamines, and enhance vasopressor responsiveness. In addition, recent evidence suggests that thiamine may be neuroprotective in severe shock states.

Specific Aims of the Study:

The aim of this study is to determine the effect of the combination of intravenous vitamin C, hydrocortisone and thiamine on the clinical course and outcome of patients with septic shock.

Study Design:

This study will be performed at 4 tertiary Greek Intensive Care Units (ICUs). All patients admitted to any ICU of the participating hospitals with the primary diagnosis of severe sepsis or septic shock will be screened for inclusion. The diagnosis of septic shock will be based on recent consensus criteria.

ICU management protocol:

All septic patients enrolled in this study will be managed by a standardized approach which will comprise:

i. Empirical treatment with broad spectrum antibiotics, which will be subsequently deescalated according to microbiological data and clinical improvement ii. A conservative strategy of fluid and vasopressor management. iii. A lung-protective ventilation strategy. iv. Limited use of sedative agents (dexmedetomidine will be the preferred agent) v. Enteral nutrition with a whey-based formula using an intermittent bolus protocol which will preferrably be started within 24 hours of ICU admission.

vi. Prophylaxis against deep venous thrombosis prophylaxis with both enoxaparin (or heparin in patients with a calculated creatinine clearance < 30ml/min) and sequential compression.

vii. Permissive hyperglycemia (blood glucose of 150-200 mg/dL).

Vitamin C, Hydrocortisone and Thiamine dosing protocol and randomization

This is a double-blind placebo controlled study. Only the pharmacist will be aware of the treatment allocation. Patients will be randomized to receive either vitamin C/hydrocortisone or placebo plus placebo using a random number table provided to the dispensing pharmacists. Each patient will be allocated a unique participant ID which will be linked to the randomization sequence. Only the dispensing pharmacists will have a record of the participant ID and randomization sequence. The vitamin C/placebo and hydrocortisone/placebo will be formulated as follows:

Vitamin C: 1500 mg of vitamin C will be dissolved in a 50 or 100 mL bag of normal saline and will be infused over 1 hour. The dosing schedule will be 1500 mg every 6 hours for 4 days or until discharge from the ICU.

Vitamin C placebo will consist of an identical bag of 50 or 100 mL normal saline (but with no vitamin C) and will be labeled vitamin C. Placebo will be infused over 1 hour as per the infusion instructions of the active vitamin.

Hydrocortisone: Patients will be treated with hydrocortisone 50mg IV q 6 hourly for 4 days or until ICU discharge.

Optional dosing strategy: Hydrocortisone 50 mg bolus, followed by a 24-hour continuous infusion of 200 mg (in 50 or 100 ml normal saline) for 4 days.

Hydrocortisone placebo will be provided as an identical syringe/50 or 100 mL bag of normal saline.

Thiamine: As a high percentage of septic patients have been shown to be thiamine deficient, patients will receive intravenous thiamine 200mg q 12 hourly for 4 days or until ICU discharge. Thiamine is also a cofactor for the metabolism of oxalate (a byproduct of vitamin C metabolism), with thiamine deficiency increasing oxalate levels. To simplify the study, both the intervention and control group will receive thiamine.

ELIGIBILITY:
Inclusion Criteria:

* i. Diagnosis of septic shock within 12 hours of admission to the ICU

Exclusion Criteria:

* i. Age < 18 years ii. Pregnant iii. Patients with an end-stage underlying disease who are unlikely to survive to hospital discharge iv. Patients with acquired immunodeficiency syndrome and a CD4 count of < 50 per microliter v. Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency. vi. Patients with septic shock transferred from another hospital vii. Patients with septic shock for more than 12 hours viii. Patients who require off-label treatment with corticosteroids for an indication other than sepsis ix. Lack of written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | 90 days
  Death before hospital discharge

SECONDARY OUTCOMES:
60-day mortality | 60 days
  Death before day 60 post-randomization
28-day mortality | 28 days
  Death before day 28 post-randomization
Procalcitonin (PCT) clearance . | 4 days
  Will be defined as baseline PCT minus PCT at 96 hours post-randomization, divided by the initial PCT and multiplied by 100
Delta Sequential Organ Failure Assessment (SOFA) score | 4 days
  Will be defined as the initial Sequential Organ Failure Assessment (SOFA) score minus the day 4 post-randomization SOFA score.
  The SOFA score is the sum of 6 subscores that range from 0 to 4 and provide an assessment of the function of the following organs/systems: Respiratory, Nervous, Cardiovascular, Liver, Coagulation, and Renal. An increasing SOFA subscore (from 0 to 1, 2, 3, and 4) indicates worsening function culminating into failure of the corresponding organ/system. The maximum possible total SOFA score equals to 24. A SOFA score of 15 or more has been previously associated with a mortality rate of more than 90%.
Neurologic failure-free days (defined as daily follow-up Glasgow Coma Score >9) within the first 28 days of follow-up | 28 days
  Will be defined as the number of days with a (daily) follow-up Glasgow Coma Score >9 within the first 28 days of follow-up
Intensive Care Unit (ICU) mortality | 90 days
  Death before ICU discharge
ICU free days to day 28. | 28 days
  Will be defined as the number of days alive and out of the ICU until follow-up day 28
ICU length of stay | 90 days
  Duration of the need for intensive care after randomization
Hospital length of stay | 90 days
  Duration of hospitalization after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Kotanidou, MD, PHD, Professor, Principal Investigator — National and Kapodestrian University of Athens, Greece; Spyros D Mentzelopoulos, MD, PHD, Associate Professor, Principal Investigator — National and Kapodestrian University of Athens, Greece; Stylianos Orfanos, MD, PHD, Professor, Study Director — National and Kapodestrian University of Athens, Greece; Spyros G Zakynthinos, MD, PHD, Professor, Study Chair — National and Kapodestrian University of Athens, Greece
Locations (2):
- Greece (2):
  - Evaggelismos General Hospital, Athens, Attica
  - General Hospital of Nikaia Saint Panteleimon, Piraeus, Attica

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan

REFERENCES:
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189